CLINICAL TRIAL: NCT03698084
Title: REspiratory Syncytial Virus Consortium in EUrope (RESCEU) Study: Defining the Burden of Respiratory Syncytial Virus (RSV) Disease.
Brief Title: RESCEU: Defining the Burden of RSV Disease
Status: Active, not recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/01
Record Dates: First submitted 2017-09-19; First posted 2018-10-05 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Respiratory Syncytial Virus Infections; RSV Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood; transcriptomics, serum, whole blood Nasopharyngeal swabs; PCR, virology, microbiome Stool; microbiome Urine; metabolome
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active: 200 infants enrolled; family demographics collected and samples at day 5 (venepuncture, nasopharyngeal swab, urine and stool), actively followed up through their first RSV season for signs of respiratory symptoms. If respiratory symptoms are due to RSV infection (by point of care testing) samples as taken at day 5 are repeated at time of infection and again 7 weeks later. Annual questionnaire enquiring into respiratory illness, hospitalisations and family health and health quality of life, for up to 3 years.
  Interventions: Procedure: venepuncture; Procedure: nasopharyngeal swab
- Passive: 1800 infants enrolled; family demographics collected. Questionnaire follow up at 1 year of age enquiring into respiratory illness, hospitalisations and family health and health quality of life. If infant was hospitalised in first year of life, follow up will continue for up to 3 years.

INTERVENTIONS:
Procedure: venepuncture — sample collection for analysis
  Groups: Active
Procedure: nasopharyngeal swab — sample collection for analysis
  Groups: Active

SUMMARY:
This observational study will determine the burden of RSV disease in at least 2000 healthy infants over 6 years until November 2026. The study will determine the incidence of acute respiratory tract infection (ARTI) associated with RSV, of medically attended ARTI and RSV related hospitalisation.

Mortality (RSV associated and all-cause) through all RSV seasons and the health care costs, resource use and Health Related Quality of Life will also be determined. The study also aims to determine important risk factors for RSV infection (by severity and healthcare utilisation.

DETAILED DESCRIPTION:
Infants will be recruited into one of two cohorts:

Passive (around 1800 participants) - Demographic data will be collected at inclusion and a parental questionnaire at one year of age. Infants admitted to a hospital with an acute respiratory tract illness will be followed up to the age of 3 years or 6 years with additional consent.

Active (around 200 participants) - Demographic data, parental questionnaire and the following samples will be collected at inclusion; blood, nasopharyngeal swabs, urine and stool. During the infants first RSV season (Oct - May) weekly phone contact will monitor respiratory symptoms. Infants with respiratory symptoms associated with RSV (confirmed by point of care testing) will have further samples of blood, nasopharyngeal swabs, urine and stool collected at the time of infection and 7 weeks later. Infants in the active cohort will be followed up for up to 3 years or 6 years with additional consent.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children, gestation age at least 37+0 weeks, born at participating centres.
* Written informed consent obtained from the mother.
* Parents able and willing to adhere to protocol-specified procedures (active cohort).

Exclusion Criteria:

* Major congenital defects or serious chronic illness (i.e. severe congenital heart and/or lung disease, genetic, immunologic and/or metabolic disorder).
* Gestational age of less than 37+0 weeks.
* Acute severe medical condition at moment of sampling (e.g. sepsis, severe asphyxia, for which the child is admitted to the hospital).
* Child in care.
* Parents not able to understand and communicate in the local language.
* Living outside catchment area of study sites.
* Mother vaccinated against RSV during pregnancy (by parental report).

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Healthy children, gestation age at least 37+0 weeks, born at participating centres and recruited within the first week of life.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-09-05 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of RSV associated Acute Respiratory Tract infections (ARTI) during the first year of life, to include the number of medically attended ARTI (MA-ARTI) and hospital admissions related to RSV. | Year 1
  RSV associated ARTI confirmed on nasopharyngeal swabs during home visits for all ARTI episodes during the RSV season, for testing using a RSV POC (Point of Care) test and reverse transcription-polymerase chain reaction (RT-PCR).
  Participants will be screened for hospital admission for respiratory symptoms by parental questionnaire at age 1 year. If positive, RSV will be confirmed by accessing hospital records.
  Medically attended RSV infection is defined as any medical care for RSV infection (defined as above)
The relationship between infant RSV infection of different severity and school age asthma | Year 4
  Symptoms of asthma, diagnosis and use of asthma medication will be measured by parental questionnaire/medical records.
The relationship between infant RSV infection of different severity and school age asthma | Year 5
  Symptoms of asthma, diagnosis and use of asthma medication will be measured by parental questionnaire/medical records.
The relationship between infant RSV infection of different severity and school age asthma | Year 6
  Symptoms of asthma, diagnosis and use of asthma medication will be measured by parental questionnaire/medical records.

SECONDARY OUTCOMES:
Wheeze symptoms up to 3 years of age following RSV infection of different severity | Year 1 - 3
  Parent reported wheeze and doctor diagnosis of wheeze by routine care (for active birth cohort and children of passive birth cohort admitted for ARTI).
Rate of all-cause medically attended (inpatient or outpatient) ARTI (active cohort). | Year 1
  Medically attended ARTI is defined as any medical care for a respiratory infection
RSV associated and all-cause mortality through all RSV seasons of follow up (passive and active cohorts). | Year 1 - 3
  Mortality through all RSV seasons of follow up including RSV-associated deaths and all cause deaths.
Health care costs and resource use | Year 1 - 3
  Health care utilisation for RSV-associated and all-cause medically attended (inpatient or outpatient) ARTI or respiratory events (active birth cohort).
Incidence of RSV-related secondary bacterial RTIs within 21 days after onset of RSV infection and their association with antibiotic use in hospitalized RSV ARTI patients and non-hospitalized RSV ARTI patients. | Within 21 days of RSV infection
  The incidence of RSV-associated secondary bacterial pneumonia and associated antibiotic consumption events within 21 days after onset of RSV-related symptoms.
To collect clinical samples (blood, nasopharyngeal, stool and urine) for biomarker analysis (active cohort). | Year 1
  Biomarkers associated with RSV infection in infants
Incidence rate of other respiratory pathogens (influenza, rhinovirus, human metapneumovirus, parainfluenzavirus, etc.) associated with all medically attended (inpatient or outpatient) ARTI (active cohort). | Year 1
  Additional viruses as detected by PCR testing on nasopharyngeal swab. Medically attended ARTI is defined as any medical care for a respiratory infection.
Risk factors for RSV infection (by severity and healthcare utilisation) (active and passive cohort). | Year 1 - 3
  Demographic risks factors as outlined in CRF/demographic questionnaires
The proportion of viral ARTI attributable to RSV (active cohort). | Year 1
  RSV and additional viruses as determined by PCR testing of nasopharyngeal swabs
Health Related Quality of Life in RSV-associated and all-cause medically attended ARTI patients and their families (active cohort). | Year 1-3
  Annual questionnaire to families to determine interruption of normal activities associated with RSV and all-cause medically attended ARTI (active cohort).
Risk factors for persistent wheeze at 3 and 6 years of age | Year 4,5 and 6
  Demographic and clinical parameters and outcomes from CRF/demographic questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided